CLINICAL TRIAL: NCT02938169
Title: The Effect of Lumbar Stabilization Exercise and Gait Training on Lower Back Muscles- Electromyographic(EMG) Analysis
Acronym: EMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-1604-344-004
Record Dates: First submitted 2016-10-13; First posted 2016-10-19 (Estimated); Results first posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Low Back Pain
Keywords: low back pain; exercise; electromyography
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- walking exercise group (Experimental): **walking exercise with bracing exercise
  * walking exercise: treadmill gait with tolerable gait speed
  * bracing exercise: patient is instructed as follows: "Draw your navel up towards your head and in toward your spine without moving your pelvis. Continue to breathe normally as you do this."
  Interventions: Behavioral: exercise
- stabilization exercise group (Experimental): ** stabilization exercise with bracing exercise
  * stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  * bracing exercise: patient is instructed as follows: "Draw your navel up towards your head and in toward your spine without moving your pelvis. Continue to breathe normally as you do this."
  Interventions: Behavioral: exercise
- walking and stabilization exercise group (Experimental): **walking exercise, bracing exercise with stabilization exercise
  * stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  * bracing exercise: patient is instructed as follows: "Draw your navel up towards your head and in toward your spine without moving your pelvis. Continue to breathe normally as you do this."
  * walking exercise:treadmill gait with tolerable gait speed
  Interventions: Behavioral: exercise
- flexibility exercise group (Sham Comparator): **Stretching exercise(control)
  * Only educate the flexibility exercise(stretching exercise)
  * Don't educate the walking exercise method and stabilization exercise method
  Interventions: Behavioral: exercise

INTERVENTIONS:
Behavioral: exercise — * stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  * bracing exercise: patient is instructed as follows: "Draw your navel up towards your head and in toward your spine without moving your pelvis. Continue to breathe normally as you do this."
  * walking exercise: treadmill gait with tolerable gait speed
  * flexibility exercise: stretching exercise(control)

SUMMARY:
The purpose of this study is to determine the effective exercise protocol in chronic low back pain patients.

DETAILED DESCRIPTION:
* Design: Prospective study
* Setting: hospital rehabilitation department
* Intervention: Participants are randomly assigned 4 different exercise group: flexibility exercise, bracing exercise + stabilization exercise group, bracing exercise+ walking exercise group and bracing+ walking + stabilization exercise group
* Main outcome measures: Numeric rating scale(NRS), Oswestry disability index Peak torque of lumbar extensor by surface electromyography Time duration of capability of maintenance the posture

ELIGIBILITY:
* Inclusion Criteria:

  * Age>20
  * Who suffered low back pain more than 3 months.
* Exclusion Criteria:

  * Pregnancy
  * Under 20-year-old
  * Who have significant neurologic deficit
  * Who experienced spine operation
  * Who cannot walking

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05; Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juseok Ryu, MD, PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Kyungji-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee HI, Lee ST, Kim M, Ryu JS. Sex differences in predicting chronicity of low-back pain after acute trauma using lumbar muscle area. Am J Phys Med Rehabil. 2015 Feb;94(2):123-30. doi: 10.1097/PHM.0000000000000149. PMID 25122093

RESULTS

PARTICIPANT FLOW:
Groups:
- Walking Exercise Group: **walking exercise
  •walking exercise: treadmill gait with tolerable gait speed
- Stabilization Exercise Group: ** stabilization exercise
  •stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
- Walking and Stabilization Exercise Group: **walking exercise with stabilization exercise
  * stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  * walking exercise:treadmill gait with tolerable gait speed
Period: Overall Study
Arm/Group | Walking Exercise Group | Stabilization Exercise Group | Walking and Stabilization Exercise Group | Flexibility Exercise Group
Started | 15 | 15 | 15 | 15
Completed | 13 | 13 | 10 | 12
Not Completed | 2 | 2 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Walking Exercise Group | Stabilization Exercise Group | Walking and Stabilization Exercise Group | Flexibility Exercise Group | Total
Number analyzed (Participants) | 13 | 10 | 12 | 13 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.15 (13.89) | 57.40 (15.88) | 54.75 (14.98) | 53.54 (15.69) | 54.81 (14.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 4 | 5 | 15
  Male | 11 | 6 | 8 | 8 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 13 | 10 | 12 | 13 | 48
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 13 | 10 | 12 | 13 | 48

OUTCOME MEASURES:

1. Primary Outcome: Low Back Pain at Resting Status
Description: numerical rating scale (NRS) (Unit: Point) Subjects indicate pain in columns 0 (no pain) to 100 (uncontrollable pain).
Time Frame: Baseline Pre-Exercise and 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Stabilization Exercise Group: ** stabilization exercise
  * stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  * bracing exercise: patient is instructed as follows: "Draw your navel up towards your head and in toward your spine without moving your pelvis. Continue to breathe normally as you do this."
  exercise: -stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  -bracing exercise: patient is instructed as follows: "Draw your navel up towards your head and in toward your spine without moving your pelvis. Continue to breathe normally as
- Walking and Stabilization Exercise Group: **walking exercise with stabilization exercise
  * stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  * walking exercise:treadmill gait with tolerable gait speed
  exercise: -stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  -bracing exercise: patient is instructed as follows: "Draw your navel up towards your head and i
- Flexibility Exercise Group: **Stretching exercise(control)
  * Only educate the flexibility exercise(stretching exercise)
  * Don't educate the walking exercise method and stabilization exercise method
  exercise: -stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  * bracing exercise: patient is instructed as follows: "Draw your navel up towards your head and in toward your spine without moving your pelvis. Continue to breathe normally as you do this."
  * walking exercise: treadmill gait with tolerable gait speed
  * flexibility exercise: stretching exercise(control)
Arm/Group | Walking Exercise Group | Stabilization Exercise Group | Walking and Stabilization Exercise Group | Flexibility Exercise Group
Number analyzed (Participants) | 13 | 10 | 12 | 13
score on a scale
  Pre-exercise | 30.58 (20.92) | 37.50 (21.76) | 30.00 (30.38) | 41.92 (23.32)
  After 6 weeks | 25.00 (20.10) | 24.25 (20.21) | 18.33 (20.93) | 27.89 (18.54)

2. Primary Outcome: Disability for Low Back Pain
Description: Oswestry disability index(ODI) (Unit: Point) The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.[
Time Frame: Baseline Pre-Exercise and 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Walking Exercise Group: **walking exercise with bracing exercise
  * walking exercise: treadmill gait with tolerable gait speed
  * bracing exercise: patient is instructed as follows: "Draw your navel up towards your head and in toward your spine without moving your pelvis. Continue to breathe normally as you do this."
  exercise: -stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  * bracing exercise: patient is instructed as follows: "Draw your navel up towards your head and in toward your spine without moving your pelvis. Continue to breathe normally as you do this."
  * walking exercise: treadmill gait with tolerable gait speed
  * flexibility exercise: stretching exercise(control)
- Stabilization Exercise Group: ** stabilization exercise with bracing exercise
  •stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  exercise: -stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  -bracing exercise: patient is instructed as follows: "Draw your navel up towards your head and in toward your spine without moving your pelvis. Continue to
- Walking and Stabilization Exercise Group: **walking exercise, bracing exercise with stabilization exercise
  * stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  * walking exercise:treadmill gait with tolerable gait speed
  exercise: -stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  -bracing exercise: patient is instructed as follows: "Draw your navel up towar
Arm/Group | Walking Exercise Group | Stabilization Exercise Group | Walking and Stabilization Exercise Group | Flexibility Exercise Group
Number analyzed (Participants) | 13 | 10 | 12 | 13
score on a scale
  Pre-exercise | 28.1 (12.8) | 31.4 (13.2) | 30.4 (12.9) | 38.0 (21.1)
  After 6 weeks | 22.5 (7.4) | 25.3 (9.9) | 24.9 (12.3) | 31.9 (18.6)

3. Primary Outcome: Visual Analog Scale of Low Back Pain During Rest
Description: visual analog scale of low back pain during resting status at 0 week and 6 week Record 'no pain' on the left side of the line as 'unpaid pain' on the right side and indicate the degree of pain in the subject(0 to 100) 0 is equated with 'no pain' and 100 is 'unpaid pain'
Time Frame: 0 week to 6weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Stabilization Exercise Group: ** stabilization exercise with bracing exercise
  •stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
- Walking and Stabilization Exercise Group: **walking exercise, bracing exercise with stabilization exercise
  * stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  * walking exercise:treadmill gait with tolerable gait speed
Arm/Group | Walking Exercise Group | Stabilization Exercise Group | Walking and Stabilization Exercise Group | Flexibility Exercise Group
Number analyzed (Participants) | 13 | 10 | 12 | 13
score on a scale | 20.00 (17.58) | 22.50 (23.72) | 20.83 (26.44) | 32.50 (21.79)

4. Secondary Outcome: Muscle Strength(Endurance)
Description: endurances of specific posture (sec) (supine, side-lying and prone)
Time Frame: Baseline Pre-Exercise and 6 weeks
Measure: Mean (Standard Deviation); unit: second
Groups:
- Stabilization Exercise Group: ** stabilization exercise with bracing exercise
  •stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  exercise: -stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  * bracing exercise: patient is instructed as follows: "Draw your navel up towards your head and in toward your spine without moving your pelvis. Continue to breathe normally as you do this."
  * walking exercise: treadmill gait with tolerable gait speed
  * flexibility exercise: stretching exercise(control)
Arm/Group | Walking Exercise Group | Stabilization Exercise Group | Walking and Stabilization Exercise Group | Flexibility Exercise Group
Number analyzed (Participants) | 13 | 10 | 12 | 13
second
  Pre-exercise | 29.86 (13.53) | 51.45 (12.40) | 35.14 (20.64) | 41.25 (15.31)
  After 6 weeks | 43.30 (18.83) | 45.06 (14.01) | 43.79 (17.81) | 50.06 (16.65)

5. Secondary Outcome: Depression Scale
Description: Beck depression inventory consisted of 21 questions about how the subject has been feeling in the last week. Each question had a set of four possible responses, ranging in intensity(0 is weak and 3 is severe). When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity. The standard cut-off scores were as follows 0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression. The total score is 63, higher total scores indicate more severe depressive symptoms.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Walking and Stabilization Exercise Group: **walking exercise, bracing exercise with stabilization exercise
  * stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  * walking exercise:treadmill gait with tolerable gait speed
  exercise: -stabilization exercise: Lumbar stabilization is a multi-component program and involves education/training, strength, flexibility, and endurance. It is generally used during all phases of a back pain episode and may be prescribed after a thorough evaluation of the patient's specific condition.
  * bracing exercise: patient is instructed as follows: "Draw your navel up towards your head and in toward your spine without moving your pelvis. Continue to breathe normally as you do this."
  * walking exercise: treadmill gait with tolerable gait speed
Arm/Group | Walking Exercise Group | Stabilization Exercise Group | Walking and Stabilization Exercise Group | Flexibility Exercise Group
Number analyzed (Participants) | 13 | 10 | 12 | 13
score on a scale
  Pre-exercise | 10.5 (7.3) | 7.2 (4.8) | 13.3 (11.9) | 12.3 (7.6)
  After 6 weeks | 8.6 (7.1) | 5.3 (6.2) | 10.7 (9.2) | 10.8 (6.7)

ADVERSE EVENTS:
Time Frame: 12weeks
Description: This study did not exceed the minimal risk, so a data safety monitoring plan would not be needed.
  There were no adverse event.
Arm/Group | Walking Exercise Group | Stabilization Exercise Group | Walking and Stabilization Exercise Group | Flexibility Exercise Group
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10 | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/10 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/10 | 0/12 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT02938169/Prot_SAP_000.pdf